CLINICAL TRIAL: NCT02032433
Title: CTN-0051: Extended-Release Naltrexone vs. Buprenorphine for Opioid Treatment
Brief Title: Extended-Release Naltrexone vs. Buprenorphine for Opioid Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); The Emmes Company, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-03133; UG1DA013035 (NIH)
Record Dates: First submitted 2013-12-30; First posted 2014-01-10 (Estimated); Results first posted 2018-01-19 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-07

CONDITIONS: Opioid Use Disorder
Keywords: extended-release naltrexone (Vivitrol); buprenorphine-naloxone (Suboxone); comparative effective; relapse prevention
MeSH Terms: conditions — Opioid-Related Disorders | interventions — vivitrol; Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Extended-Release Naltrexone (Active Comparator): Extended-Release Naltrexone (Vivitrol)
  Interventions: Drug: Extended-Release Naltrexone
- Buprenorphine-Naloxone (Active Comparator): Buprenorphine-Naloxone (Suboxone)
  Interventions: Drug: Buprenorphine-Naloxone

INTERVENTIONS:
Drug: Extended-Release Naltrexone — Extended-Release Naltrexone (Vivitrol®)
  Other Names: Vivitrol®
  Arms: Extended-Release Naltrexone
Drug: Buprenorphine-Naloxone — Buprenorphine-Naloxone (Suboxone®)
  Other Names: Suboxone®
  Arms: Buprenorphine-Naloxone

SUMMARY:
CTN-0051 assesses the comparative effectiveness of extended release injectable naltrexone (XR-NTX, Vivitrol®), an opioid antagonist recently approved and indicated for the prevention of relapse to opioid dependence, versus buprenorphine-naloxone (BUP-NX, Suboxone®), a high affinity partial agonist indicated for maintenance treatment of opioid dependence, as pharmacotherapeutic aids to recovery.

The study is conducted in 8 NIDA Clinical Trials Network affiliated community based treatment programs. Up to 600 eligible participants will be randomized to treatment with XR-NTX or BUP-NX for 24 weeks (sufficient to include 350 participants who are randomized more than 72 hours after their last opioid).

The primary goal of the study is to estimate the difference, if one exists, between XR-NTX and BUP-NX in the distribution of the time to relapse (i.e.., loss of persistent abstinence) during the 6-month trial. Secondary objectives are to: (1) compare outcome on XR-NTX versus BUP-NX across a range of clinical safety and secondary efficacy domains, and (2) explore demographic and, clinical, and genetic predictors of successful treatment and moderators of differential effectiveness (i.e., what variables may help clinicians choose which of these treatments is best for a given patient).), and (3) collect a limited dataset to permit analyses of economic costs and benefits of the two treatments.

DETAILED DESCRIPTION:
For opioid-dependent patients in the U.S. and most of the rest of the world, detoxification or detoxification followed by short term residential treatment, with the goal of achieving long-term abstinence from opioid misuse is a mainstay of treatment. Nonetheless, the majority of patients treated in this way will relapse to opioid misuse, leading to a costly and ineffectual cycle of readmission for repeated detoxifications.

The overarching goal of CTN-0051 is to foster adoption of new relapse-prevention pharmacotherapies in community-based treatment programs (CTPs) where these could have a substantial public health impact. To this end CTN-0051 assesses the comparative effectiveness of extended release injectable naltrexone (XR-NTX, Vivitrol®), an opioid antagonist recently approved and indicated for the prevention of relapse to opioid dependence, versus buprenorphine-naloxone (BUP-NX, Suboxone®), a high affinity partial agonist indicated for maintenance treatment of opioid dependence, as pharmacotherapeutic aids to recovery.

The study is conducted in 8 CTN-affiliated CTPs that provide or partner with detoxification services (inpatient/residential) which have the capacity to maintain participants opioid-free for approximately 3-7 days, have the capacity to provide medication-assisted therapy, and can provide a minimum of one group or individual counseling session per week during the 24-week treatment period. Up to 600 eligible participants will be randomized to treatment with XR-NTX or BUP-NX for 24 weeks (sufficient to include 350 participants who are randomized more than 72 hours after their last opioid). To maximize generalizability, the point of randomization is flexible, from shortly after program admission until just prior to program discharge. A data analysis modification (assessment of whether the early vs. late randomizers have a differential treatment effect and if so, time to relapse will be estimated for early and late randomizers separately) will occur if differential treatment initiation is a problem for cases randomized prior to completing detoxification (i.e., significantly fewer early randomizers are able to complete detoxification and XR-NTX induction).

The primary goal of the study is to estimate the difference, if one exists, between XR-NTX and BUP-NX in the distribution of the time to relapse (i.e., loss of persistent abstinence) during the 6-month trial. The primary outcome measure will be the time to the event, with the event called relapse. Secondary objectives are to: (1) compare outcome on XR-NTX versus BUP-NX across a range of clinical safety and secondary efficacy domains, and (2) explore demographic and, clinical, and genetic predictors of successful treatment and moderators of differential effectiveness (i.e., what variables may help clinicians choose which of these treatments is best for a given patient), and (3) collect a limited dataset to permit analyses of economic costs and benefits of the two treatments.

Toward the end of the 24-week treatment period, participants are referred for follow-up care in the community (which could include pharmacotherapy if desired and available), and follow-up outcomes are assessed at week 28 and week 36 after randomization. For participants receiving BUP-NX, who do not wish to continue, or for whom community resources are not available, the study provides a two-week BUP-NX taper.

In an ancillary genetics study we plan to study functional variants in three genes (OPRM1, OPRK1 and PDYN), known to affect the dynamic response to opioid receptor ligands. These variants will be evaluated in CTN-0051 for their contribution to treatment retention, abstinence, and depression. Blood collection for DNA extraction will occur at the same time that blood is collected for medical safety and liver function evaluation, precluding the need for an additional needle-stick. Coded blood samples for the genetics studies will be sent to the NIDA Center for Genetics Repository.

ELIGIBILITY:
Inclusion Criteria

* Male or female
* 18 years of age and older
* Meet DSM-5 criteria for opioid-use disorder (heroin and/or prescription opioids)
* Have used opioids other than as specifically prescribed within thirty days prior to consent
* Seeking treatment for opioid dependence and willing to accept "agonist-based" or "antagonist-based" therapy
* In good-enough general health, as determined by the study physician on the basis of medical history, review of systems, physical exam and laboratory assessments, to permit treatment with XR-NTX or BUP-NX
* Able to provide written informed consent
* Able to speak English sufficiently to understand the study procedures and provide written informed consent to participate in the study
* If female of childbearing potential, be willing to practice an effective method of birth control for the duration of participation in the study

Exclusion Criteria

* Serious medical, psychiatric or substance use disorder that, in the opinion of the study physician, would make study participation hazardous to the participant, or compromise study findings or would prevent the participant from completing the study. Examples include:

  1. Disabling or terminal medical illness (e.g., uncompensated heart failure, cirrhosis or end-stage liver disease) as assessed by medical history, review of systems, physical exam and/or laboratory assessments;
  2. Severe, untreated or inadequately treated mental disorder (e.g., active psychosis, uncontrolled manic-depressive illness) as assessed by history and/or clinical interview;
  3. Current severe alcohol, benzodiazepine, or other depressant or sedative hypnotic use likely to require a complicated medical detoxification (routine alcohol and sedative detoxifications may be included)
* LFTs (ALT, AST) greater than 5 times upper limit of normal
* Suicidal or homicidal ideation that requires immediate attention
* Known allergy or sensitivity to buprenorphine, naloxone, naltrexone, polylactide-co-glycolide, carboxymethylcellulose, or other components of the Vivitrol® diluent
* Maintenance on methadone at doses of 30mg or greater at the time of signing consent
* Presence of pain of sufficient severity as to require ongoing pain management with opioids
* Pending legal action or other reasons that might prevent an individual from completing the study
* If female, currently pregnant or breastfeeding, or planning on conception
* Body habitus that, in the judgment of the study physician, precludes safe intramuscular injection of XR-NTX (e.g., BMI>40, excess fat tissue over the buttocks, emaciation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 570 (Actual)
Dates: Start 2014-01-29 (Actual); Primary Completion 2017-01-25 (Actual); Study Completion 2017-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Rotrosen, MD, Principal Investigator — NYU Langone Health
Locations (8):
- United States (8):
  - Tarzana Treatment Centers, Tarzana, California
  - Gateway Community Services, Inc., Jacksonville, Florida
  - Avery Road Treatment Center, Rockville, Maryland
  - Stanley Street Treatment and Resources, Fall River, Massachusetts
  - Turquoise Lodge Hospital, Albuquerque, New Mexico
  - Bellevue Hospital Center, New York, New York
  - Maryhaven, Columbus, Ohio
  - Evergreen Treatment Services, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
Data from this study will be available to researchers on the website, http://datashare.nida.nih.gov/ after the study is complete and the data analyzed. This website will not include information that can identify individual study participants.

REFERENCES:
- [Derived] Kornor H, Lobmaier PPK, Kunoe N. Sustained-release naltrexone for opioid dependence. Cochrane Database Syst Rev. 2025 May 9;5(5):CD006140. doi: 10.1002/14651858.CD006140.pub3. PMID 40342086
- [Derived] Brandt L, Odom GJ, Hu MC, Castro C, Balise RR; CTN-0094 Team. Empirically contrasting urine drug screening-based opioid use disorder treatment outcome definitions. Addiction. 2024 Jul;119(7):1289-1300. doi: 10.1111/add.16494. Epub 2024 Apr 14. PMID 38616571
- [Derived] Foot C, Korthuis PT, Tsui JI, Luo SX, Chan B, Cook RR. Associations between stimulant use and return to illicit opioid use following initiation onto medication for opioid use disorder. Addiction. 2024 Jan;119(1):149-157. doi: 10.1111/add.16334. Epub 2023 Sep 15. PMID 37712113
- [Derived] Nielsen S, Tse WC, Larance B. Opioid agonist treatment for people who are dependent on pharmaceutical opioids. Cochrane Database Syst Rev. 2022 Sep 5;9(9):CD011117. doi: 10.1002/14651858.CD011117.pub3. PMID 36063082
- [Derived] Tsui JI, Campbell ANC, Pavlicova M, Choo TH, Lee JD, Cook RR, Shulman M, Nunes EV, Rotrosen J. Methamphetamine/amphetamine use over time among persons with opioid use disorders treated with buprenorphine/naloxone versus extended-release naltrexone. Drug Alcohol Depend. 2022 Jul 1;236:109469. doi: 10.1016/j.drugalcdep.2022.109469. Epub 2022 Apr 21. PMID 35605529
- [Derived] Jelovac A, McLoughlin DM. Twelve-Month Outcomes for Remitters Following Electroconvulsive Therapy for Depression. J Clin Psychiatry. 2022 Apr 18;83(3):21lr14371. doi: 10.4088/JCP.21lr14371. No abstract available. PMID 35452195
- [Derived] Na PJ, Scodes J, Fishman M, Rotrosen J, Nunes EV. Co-occurring Depression and Suicidal Ideation in Opioid Use Disorder: Prevalence and Response During Treatment With Buprenorphine-Naloxone and Injection Naltrexone. J Clin Psychiatry. 2022 Apr 18;83(3):21m14140. doi: 10.4088/JCP.21m14140. PMID 35452194
- [Derived] Rudolph KE, Shulman M, Fishman M, Diaz I, Rotrosen J, Nunes EV. Association between dynamic dose increases of buprenorphine for treatment of opioid use disorder and risk of relapse. Addiction. 2022 Mar;117(3):637-645. doi: 10.1111/add.15654. Epub 2021 Oct 1. PMID 34338389
- [Derived] Nunes EV Jr, Scodes JM, Pavlicova M, Lee JD, Novo P, Campbell ANC, Rotrosen J. Sublingual Buprenorphine-Naloxone Compared With Injection Naltrexone for Opioid Use Disorder: Potential Utility of Patient Characteristics in Guiding Choice of Treatment. Am J Psychiatry. 2021 Jul;178(7):660-671. doi: 10.1176/appi.ajp.2020.20060816. Epub 2021 Jun 25. PMID 34170188
- [Derived] Fishman M, Wenzel K, Scodes J, Pavlicova M, Campbell ANC, Rotrosen J, Nunes E. Examination of Correlates of OUD Outcomes in Young Adults: Secondary Analysis From the XBOT Trial. Am J Addict. 2021 Sep;30(5):433-444. doi: 10.1111/ajad.13176. Epub 2021 Jun 1. PMID 34075644
- [Derived] Shulman M, Choo TH, Scodes J, Pavlicova M, Wai J, Haenlein P, Tofighi B, Campbell ANC, Lee JD, Rotrosen J, Nunes EV. Association between methadone or buprenorphine use during medically supervised opioid withdrawal and extended-release injectable naltrexone induction failure. J Subst Abuse Treat. 2021 May;124:108292. doi: 10.1016/j.jsat.2021.108292. Epub 2021 Jan 16. PMID 33771287
- [Derived] Lee JD, Nunes EV Jr, Novo P, Bachrach K, Bailey GL, Bhatt S, Farkas S, Fishman M, Gauthier P, Hodgkins CC, King J, Lindblad R, Liu D, Matthews AG, May J, Peavy KM, Ross S, Salazar D, Schkolnik P, Shmueli-Blumberg D, Stablein D, Subramaniam G, Rotrosen J. Comparative effectiveness of extended-release naltrexone versus buprenorphine-naloxone for opioid relapse prevention (X:BOT): a multicentre, open-label, randomised controlled trial. Lancet. 2018 Jan 27;391(10118):309-318. doi: 10.1016/S0140-6736(17)32812-X. Epub 2017 Nov 14. PMID 29150198
- [Derived] Lee JD, Nunes EV, Mpa PN, Bailey GL, Brigham GS, Cohen AJ, Fishman M, Ling W, Lindblad R, Shmueli-Blumberg D, Stablein D, May J, Salazar D, Liu D, Rotrosen J. NIDA Clinical Trials Network CTN-0051, Extended-Release Naltrexone vs. Buprenorphine for Opioid Treatment (X:BOT): Study design and rationale. Contemp Clin Trials. 2016 Sep;50:253-64. doi: 10.1016/j.cct.2016.08.004. Epub 2016 Aug 10. PMID 27521809

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Extended-Release Naltrexone | Buprenorphine-Naloxone
Started | 283 | 287
Completed | 205 | 225
Not Completed | 78 | 62

BASELINE CHARACTERISTICS:
Population: Adults with DSM-5 OUD with non prescribed opioid use in the past 30 days.
Groups:
- Total: Total of all reporting groups
Arm/Group | Extended-Release Naltrexone | Buprenorphine-Naloxone | Total
Number analyzed (Participants) | 283 | 287 | 570
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.0 (9.5) | 33.7 (9.8) | 33.9 (9.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 81 | 169
  Male | 195 | 206 | 401
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 45 | 54 | 99
  Not Hispanic or Latino | 238 | 233 | 471
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 8 | 1 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 29 | 28 | 57
  White | 206 | 215 | 421
  More than one race | 18 | 14 | 32
  Unknown or Not Reported | 20 | 27 | 47
Randomization status [Count of Participants; unit: Participants]
  Early randomization | 107 | 110 | 217
  Late randomization | 176 | 177 | 353

OUTCOME MEASURES:

1. Primary Outcome: Time to Relapse (Intent to Treat Population)
Description: Relapse occurs if the participant is using any non-protocol prescribed opioids regularly starting at day 21 post-randomization or thereafter. Operationally, relapse is defined as either: (a) four consecutive opioid use weeks, or (b) seven consecutive days of use by self-report. A use week is defined as any week during which a participant self-reports at least one day of use during that week, provides a urine sample positive for non-protocol opioids, or fails to provide a urine sample. Self-report of opioid (heroin or prescription opioids) and other substance use is ascertained at each weekly study visit using the Timeline Follow-Back for each day leading back to the previous visit. Urine is collected at each study visit and tested for opioids. A missed UDS counts as a use week.
Time Frame: Weeks 3-24
Population: Intention to treat.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Extended-Release Naltrexone | Buprenorphine-Naloxone
Number analyzed (Participants) | 283 | 287
weeks | 8.4 [3.0 to 23.4] | 14.4 [5.1 to 23.4]

2. Primary Outcome: Time to Relapse (Per Protocol Population)
Description: as for outcome 1
Time Frame: Weeks 3-24
Population: Per protocol population (those successfully inducted onto medication)
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Extended-Release Naltrexone | Buprenorphine-Naloxone
Number analyzed (Participants) | 204 | 270
weeks | 20.4 [5.4 to 23.4] | 15.2 [5.7 to 23.4]

3. Secondary Outcome: Number Successfully Inducted Onto Assigned Study Medication
Description: Binary Y/N assessment of whether the participant was or was not able to initiate their assigned study medication.
Time Frame: Weeks 0-24
Population: Intent to treat
Measure: Number; unit: participants
Arm/Group | Extended-Release Naltrexone | Buprenorphine-Naloxone
Number analyzed (Participants) | 283 | 287
participants | 204 | 270

4. Secondary Outcome: Adverse Events Related to Study Medications
Description: Adverse events reported by participants and assessed by clinical staff for relatedness to study medication. These determinations were reviewed by the study medical monitor.
Time Frame: Weeks 0-36
Population: These are treatment emergent adverse events. Treatment emergence is defined as any adverse events that occurred after the study day of induction for those participants inducted onto study medication.
Measure: Number; unit: events
Arm/Group | Extended-Release Naltrexone | Buprenorphine-Naloxone
Number analyzed (Participants) | 204 | 270
events | 115 | 113

5. Secondary Outcome: Opioid Abstinence Over Time While on Study Medication (Subjective)
Description: Self report of opioid use by participants using the TLFB. At each visit, the TLFB was completed for dates going back to the last participant encounter.
Time Frame: Weeks 0-24
Population: per protocol
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Extended-Release Naltrexone | Buprenorphine-Naloxone
Number analyzed (Participants) | 204 | 270
days | 123 [18 to 144] | 87 [20 to 144]

6. Secondary Outcome: Alcohol Use Over Time, Drinks Per Day, Past 30 Days, W0
Description: Alcohol use over time, drinks per day, past 30 days, at week 0
Time Frame: Week 0
Measure: Mean (Standard Deviation); unit: drinks per day
Arm/Group | Extended-Release Naltrexone | Buprenorphine-Naloxone
Number analyzed (Participants) | 283 | 287
drinks per day | .8 (2.41) | 1.2 (3.75)

7. Secondary Outcome: Cigarette Smoking, W0, 10 or Less
Description: Participants average cigarettes/day, in past 4 weeks, at week 0, equals 10 or less.
Time Frame: Week 0
Measure: Count of Participants; unit: Participants
Arm/Group | Extended-Release Naltrexone | Buprenorphine-Naloxone
Number analyzed (Participants) | 283 | 287
Participants | 112 | 109

8. Secondary Outcome: Opioid Craving Over Time W0
Description: Opioid craving over time via VAS at week 0
Time Frame: Week 0
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Extended-Release Naltrexone | Buprenorphine-Naloxone
Number analyzed (Participants) | 283 | 287
score on a scale | 68.7 (30.55) | 68.8 (30.05)

9. Secondary Outcome: Score of Subacute Withdrawal Symptoms Subscale Within Hamilton Depression (HAM-D) Rating Scale
Description: The Subacute Withdrawal Symptoms Subscale consists of 6 symptoms. Classification of symptoms can be scored as: 0 - absent, 1 - doubtful or trivial, 2 - present. The total range of scores is 0 - 12, and the higher the total score the more severe the depression.
Time Frame: Week 0
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Extended-Release Naltrexone | Buprenorphine-Naloxone
Number analyzed (Participants) | 283 | 287
score on a scale | 8.6 (6.45) | 9.3 (6.63)

10. Secondary Outcome: Score of Alcohol Subscale Within Addiction Severity Index (ASI) Scale
Description: The Alcohol Subscale within ASI is one question that asks how bothered one has been by alcohol problems. The total range of the subscale is 0-4. The higher the score, the bigger the problem.
Time Frame: Week 0
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Extended-Release Naltrexone | Buprenorphine-Naloxone
Number analyzed (Participants) | 283 | 287
score on a scale | .1 (.2) | .1 (.23)

11. Secondary Outcome: Score of Sexual Behavior Subscale Within HIV Risk-Taking Behavior Scale (HRBS)
Description: The Sexual Behavior Subscale consists of 5 questions. Each question is scored from 0-5, for a total score range of 0-25. Higher scores indicate a greater degree of risk-taking behavior.
Time Frame: Week 0
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Extended-Release Naltrexone | Buprenorphine-Naloxone
Number analyzed (Participants) | 283 | 287
score on a scale | 5.5 (8.85) | 5.9 (10.46)

12. Secondary Outcome: Score on Trail Making Test Part A
Description: Trail Making Test Part A consists of 25 circles distributed over a sheet of paper. The circles are number 1-25, and the patient is asked to draw lines to connect the numbers in ascending order. The patient is instructed to connect the circles as quickly as possible, without lifting the pen or pencil from the paper. Higher scores reveal greater impairment.
Time Frame: Week 0
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Extended-Release Naltrexone | Buprenorphine-Naloxone
Number analyzed (Participants) | 283 | 287
seconds | 26.8 (11.09) | 25.8 (10.07)

13. Secondary Outcome: Opioid Abstinence Over Time While on Study Medication (Objective)
Description: A urine sample was obtained and tested for opioids at each in person visit; screening, prior to induction onto study medication, weekly through week 24 and at each of the follow up visits.
Time Frame: Weeks 0-24
Population: Per protocol
Measure: Median (Inter-Quartile Range); unit: Weeks
Arm/Group | Extended-Release Naltrexone | Buprenorphine-Naloxone
Number analyzed (Participants) | 204 | 270
Weeks | 13 [3 to 21] | 11 [3 to 20]

14. Secondary Outcome: Cigarette Smoking, W0 0
Description: Participants average cigarettes/day, in past 4 weeks, at week 0, equals none
Time Frame: Week 0
Measure: Count of Participants; unit: Participants
Arm/Group | Extended-Release Naltrexone | Buprenorphine-Naloxone
Number analyzed (Participants) | 283 | 287
Participants | 17 | 18

15. Secondary Outcome: Cigarette Smoking, W0 11-20
Description: Participants average cigarettes/day, in past 4 weeks, at week 0, equals 11-20.
Time Frame: Week 0
Measure: Count of Participants; unit: Participants
Arm/Group | Extended-Release Naltrexone | Buprenorphine-Naloxone
Number analyzed (Participants) | 283 | 287
Participants | 106 | 112

16. Secondary Outcome: Cigarette Smoking, W0 21-30
Description: Participants average cigarettes/day, in past 4 weeks, at week 0, equals 21-30
Time Frame: Week 0
Measure: Count of Participants; unit: Participants
Arm/Group | Extended-Release Naltrexone | Buprenorphine-Naloxone
Number analyzed (Participants) | 283 | 287
Participants | 18 | 21

17. Secondary Outcome: Cigarette Smoking, W0 31 or More
Description: Participants average cigarettes/day, in past 4 weeks, at week 0, equals 31 or more
Time Frame: Week 0
Measure: Count of Participants; unit: Participants
Arm/Group | Extended-Release Naltrexone | Buprenorphine-Naloxone
Number analyzed (Participants) | 283 | 287
Participants | 3 | 8

18. Secondary Outcome: Cigarette Smoking, W24 0
Description: Participants average cigarettes/day, in past 4 weeks, at week 24, equals none
Time Frame: Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Extended-Release Naltrexone | Buprenorphine-Naloxone
Number analyzed (Participants) | 283 | 287
Participants | 32 | 29

19. Secondary Outcome: Cigarette Smoking
Description: Participants average cigarettes/day, in past 4 weeks, at week 24, equals 10 or less.
Time Frame: Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Extended-Release Naltrexone | Buprenorphine-Naloxone
Number analyzed (Participants) | 283 | 287
Participants | 70 | 78

20. Secondary Outcome: Cigarette Smoking, W24 11-20
Description: Participants average cigarettes/day, in past 4 weeks, at week 24, equals 11-20.
Time Frame: Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Extended-Release Naltrexone | Buprenorphine-Naloxone
Number analyzed (Participants) | 283 | 287
Participants | 57 | 71

21. Secondary Outcome: Cigarette Smoking, W24 21-30
Description: Participants average cigarettes/day, in past 4 weeks, at week 24, equals 21-30
Time Frame: Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Extended-Release Naltrexone | Buprenorphine-Naloxone
Number analyzed (Participants) | 283 | 287
Participants | 2 | 11

22. Secondary Outcome: Cigarette Smoking, W24 31 or More
Description: Participants average cigarettes/day, in past 4 weeks, at week 24, equals 31 or more
Time Frame: Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Extended-Release Naltrexone | Buprenorphine-Naloxone
Number analyzed (Participants) | 283 | 287
Participants | 1 | 5

23. Secondary Outcome: Score on Opioid Craving Scale (OCS)
Description: OCS is a brief 3-item measure used to measure opioid craving. The scale consists of 3 items rated on a visual analogue scale (VAS) from 1-10. The total range of score is 0-30, and a higher score indicates a stronger craver / desire to use opiates.
Time Frame: Week 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Extended-Release Naltrexone | Buprenorphine-Naloxone
Number analyzed (Participants) | 283 | 287
score on a scale | 9.9 (21.54) | 9.4 (17.67)

24. Secondary Outcome: Score of Subacute Withdrawal Symptoms Subscale Within Hamilton Depression (HAM-D) Rating Scale
Description: as for outcome 9
Time Frame: Week 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Extended-Release Naltrexone | Buprenorphine-Naloxone
Number analyzed (Participants) | 283 | 287
score on a scale | 5.2 (6.53) | 4.8 (5.48)

25. Secondary Outcome: Score on Subjective Opiate Withdrawal Scale (SOWS)
Description: The SOWS is a self-administered scale for grading opioid withdrawal symptoms. It contains 16 symptoms whose intensity the patient rates on a scale of 0 (not at all) to 4 (extremely). The total range of scores is 0-64; the higher the score, the more intense the withdrawal.
Time Frame: Week 0
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Extended-Release Naltrexone | Buprenorphine-Naloxone
Number analyzed (Participants) | 283 | 287
score on a scale | 15.6 (13.38) | 15.6 (13.15)

26. Secondary Outcome: Score on Subjective Opiate Withdrawal Scale (SOWS)
Description: as for outcome 25
Time Frame: Week 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Extended-Release Naltrexone | Buprenorphine-Naloxone
Number analyzed (Participants) | 283 | 287
score on a scale | 4.5 (7.53) | 5.3 (7.49)

27. Secondary Outcome: Score of Sexual Behavior Subscale Within HIV Risk-Taking Behavior Scale (HRBS)
Description: as for outcome 11
Time Frame: Week 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Extended-Release Naltrexone | Buprenorphine-Naloxone
Number analyzed (Participants) | 283 | 287
score on a scale | 7.3 (9.37) | 6.0 (10.63)

28. Secondary Outcome: Score of Condom Use Subscale Within HIV Risk-Taking Behavior Scale (HRBS)
Description: The Sexual Behavior Subscale consists of 3 questions. Each question is scored from 0-5, for a total score range of 0-15. Higher scores indicate a greater degree of risk-taking behavior.
Time Frame: Week 0
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Extended-Release Naltrexone | Buprenorphine-Naloxone
Number analyzed (Participants) | 283 | 287
score on a scale | 3.6 (7.34) | 4.3 (10.07)

29. Secondary Outcome: Score of Condom Use Subscale Within HIV Risk-Taking Behavior Scale (HRBS)
Description: as for outcome 28
Time Frame: Week 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Extended-Release Naltrexone | Buprenorphine-Naloxone
Number analyzed (Participants) | 283 | 287
score on a scale | 4.8 (8.4) | 4.3 (10.34)

30. Secondary Outcome: Score on Trail Making Test Part A
Description: as for outcome 12
Time Frame: Week 24
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Extended-Release Naltrexone | Buprenorphine-Naloxone
Number analyzed (Participants) | 283 | 287
seconds | 21.6 (9.81) | 20.3 (7.03)

31. Secondary Outcome: Score on Trail Making Test Part B
Description: Part B consists of 25 circles distributed over a sheet of paper. In Part B, the circles include both numbers (1-13) and letters (A-L); the patient draws lines to connect the circles in an ascending pattern, by alternating between the numbers and letters. Results are reported as the number of seconds required to complete the task.
Time Frame: Week 0
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Extended-Release Naltrexone | Buprenorphine-Naloxone
Number analyzed (Participants) | 283 | 287
seconds | 79.1 (40.19) | 78.3 (40.73)

32. Secondary Outcome: Score on Trail Making Test Part B
Description: as for outcome 31
Time Frame: Week 24
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Extended-Release Naltrexone | Buprenorphine-Naloxone
Number analyzed (Participants) | 283 | 287
seconds | 61.2 (39.32) | 58.1 (33.37)

33. Secondary Outcome: Score on Word Card of Stoop Test
Description: The "word card" of the Stoop Test has the names of colors printed in black and white (100 items to be named). The patient's basic score is the total time he/she takes to utter the 100 words on the card.
Time Frame: Week 0
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Extended-Release Naltrexone | Buprenorphine-Naloxone
Number analyzed (Participants) | 283 | 287
seconds | 95.8 (16.6) | 96.4 (16.03)

34. Secondary Outcome: Score on Word Card of Stoop Test
Description: as for outcome 33
Time Frame: Week 24
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Extended-Release Naltrexone | Buprenorphine-Naloxone
Number analyzed (Participants) | 283 | 287
seconds | 103.2 (18.02) | 102.9 (19.7)

35. Secondary Outcome: Score on Color Card of Stoop Test
Description: The "color card" contains 100 patches of between 3-5 different colors. The patient's task is to utter the names of the colored patches as rapidly as possible, scanning the rows from left to right. The score is the total time (in seconds) it takes to utter the 100 colors.
Time Frame: Week 0
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Extended-Release Naltrexone | Buprenorphine-Naloxone
Number analyzed (Participants) | 283 | 287
seconds | 69.3 (13.63) | 70.5 (12.46)

36. Secondary Outcome: Score on Color Card of Stoop Test
Description: as for outcome 35
Time Frame: Week 24
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Extended-Release Naltrexone | Buprenorphine-Naloxone
Number analyzed (Participants) | 283 | 287
seconds | 75.3 (15.31) | 76.1 (14.84)

37. Secondary Outcome: Score on Color Word Card of Stoop Test
Description: The "color-word card" contains the printed names of colors, but printed in an ink of a conflicting color (e.g. the word RED might be printed in green, yellow, or blue). The patient is required to name the colors of the inks while ignoring the conflicting printed color names. The basic score is the total time (in seconds) to utter the 100 colors.
Time Frame: Week 0
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Extended-Release Naltrexone | Buprenorphine-Naloxone
Number analyzed (Participants) | 283 | 287
seconds | 41.1 (10.33) | 42.2 (9.85)

38. Secondary Outcome: Score on Color Word Card of Stoop Test
Description: as for outcome 37
Time Frame: Week 24
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Extended-Release Naltrexone | Buprenorphine-Naloxone
Number analyzed (Participants) | 283 | 287
seconds | 47.6 (12.07) | 48.8 (12.35)

39. Secondary Outcome: Score of Alcohol Subscale Within Addiction Severity Index (ASI) Scale
Description: as for outcome 10
Time Frame: Week 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Extended-Release Naltrexone | Buprenorphine-Naloxone
Number analyzed (Participants) | 283 | 287
score on a scale | .1 (.11) | 0.0 (0.11)

40. Secondary Outcome: Score of Drug Use Subscale Within Addiction Severity Index (ASI) Scale
Description: The Drug Use Subscale within ASI is one question that asks how bothered one has been by drug use problems. The total range of the subscale is 0-4. The higher the score, the bigger the problem.
Time Frame: Week 0
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Extended-Release Naltrexone | Buprenorphine-Naloxone
Number analyzed (Participants) | 283 | 287
score on a scale | 0.3 (0.08) | .3 (0.09)

41. Secondary Outcome: Score of Drug Use Subscale Within Addiction Severity Index (ASI) Scale
Description: as for outcome 40
Time Frame: Week 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Extended-Release Naltrexone | Buprenorphine-Naloxone
Number analyzed (Participants) | 283 | 287
score on a scale | .1 (.13) | .1 (.12)

42. Secondary Outcome: Score of Social Relationship Subscale Within Addiction Severity Index (ASI) Scale
Description: The Social Relationship Subscale within ASI contains 2 questions that ask how bothered one has been by family or social problems. The total range of the subscale is 0-8. The higher the score, the bigger the problem.
Time Frame: Week 0
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Extended-Release Naltrexone | Buprenorphine-Naloxone
Number analyzed (Participants) | 283 | 287
score on a scale | .3 (.25) | .3 (.24)

43. Secondary Outcome: Score of Family / Social Relationship Subscale Within Addiction Severity Index (ASI) Scale
Description: The Family / Social Relationship Subscale within ASI contains 2 questions that ask how bothered one has been by family or social problems. The total range of the subscale is 0-8. The higher the score, the bigger the problem.
Time Frame: Week 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Extended-Release Naltrexone | Buprenorphine-Naloxone
Number analyzed (Participants) | 283 | 287
score on a scale | .1 (.18) | .1 (.19)

44. Secondary Outcome: Score of Legal Status Subscale Within Addiction Severity Index (ASI) Scale
Description: The Legal Status Subscale within ASI is one question that asks how bothered one has been by legal problems. The total range of the subscale is 0-4. The higher the score, the bigger the problem.
Time Frame: Week 0
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Extended-Release Naltrexone | Buprenorphine-Naloxone
Number analyzed (Participants) | 283 | 287
score on a scale | .2 (.21) | .2 (.21)

45. Secondary Outcome: Score of Legal Status Subscale Within Addiction Severity Index (ASI) Scale
Description: as for outcome 44
Time Frame: Week 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Extended-Release Naltrexone | Buprenorphine-Naloxone
Number analyzed (Participants) | 283 | 287
score on a scale | .1 (.17) | .1 (.17)

46. Secondary Outcome: Score of Medical Status Subscale Within Addiction Severity Index (ASI) Scale
Description: The Medical Status Subscale within ASI is one question that asks how bothered one has been by medical problems. The total range of the subscale is 0-4. The higher the score, the bigger the problem.
Time Frame: Week 0
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Extended-Release Naltrexone | Buprenorphine-Naloxone
Number analyzed (Participants) | 283 | 287
score on a scale | .2 (.25) | .2 (.27)

47. Secondary Outcome: Score of Medical Status Subscale Within Addiction Severity Index (ASI) Scale
Description: as for outcome 46
Time Frame: Week 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Extended-Release Naltrexone | Buprenorphine-Naloxone
Number analyzed (Participants) | 283 | 287
score on a scale | .1 (.24) | .2 (.25)

48. Secondary Outcome: Score of Psychiatric Status Subscale Within Addiction Severity Index (ASI) Scale
Description: The Psychiatric Status Subscale within ASI is one question that asks how bothered one has been by psychiatric or emotional problems. The total range of the subscale is 0-4. The higher the score, the bigger the problem.
Time Frame: Week 0
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Extended-Release Naltrexone | Buprenorphine-Naloxone
Number analyzed (Participants) | 283 | 287
score on a scale | .3 (.22) | .3 (.22)

49. Secondary Outcome: Score of Psychiatric Status Subscale Within Addiction Severity Index (ASI) Scale
Description: as for outcome 48
Time Frame: Week 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Extended-Release Naltrexone | Buprenorphine-Naloxone
Number analyzed (Participants) | 283 | 287
score on a scale | .2 (.21) | .2 (.21)

50. Secondary Outcome: Score on EuroQOL EQ-5D Questionnaire
Description: Problems related to drug abuse is assessed through this questionnaire, which consists of 5 conditions. Each condition is scored from 0-2 for a total score range of 0-10. The higher the score, the more problems.
Time Frame: Week 0
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Extended-Release Naltrexone | Buprenorphine-Naloxone
Number analyzed (Participants) | 283 | 287
score on a scale | 6.8 (1.44) | 6.8 (1.31)

51. Secondary Outcome: Score on EuroQOL EQ-5D Questionnaire
Description: as for outcome 50
Time Frame: Week 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Extended-Release Naltrexone | Buprenorphine-Naloxone
Number analyzed (Participants) | 283 | 287
score on a scale | 5.8 (1.15) | 6.1 (1.28)

52. Secondary Outcome: Alcohol Use Over Time, Drinks Per Day
Description: Alcohol use over time, drinks per day
Time Frame: Week 24
Measure: Mean (Standard Deviation); unit: drinks per day
Arm/Group | Extended-Release Naltrexone | Buprenorphine-Naloxone
Number analyzed (Participants) | 283 | 287
drinks per day | .1 (.82) | .4 (1.57)

53. Secondary Outcome: Other Drug Use Over Time, Cannabis, W0
Description: Other drug use over time measuring cannabis at week 0
Time Frame: week 0
Measure: Count of Participants; unit: Participants
Arm/Group | Extended-Release Naltrexone | Buprenorphine-Naloxone
Number analyzed (Participants) | 283 | 287
Participants | 123 | 135

54. Secondary Outcome: Other Drug Use Over Time, Cannabis, W24
Description: Other drug use over time measuring cannabis at week 24
Time Frame: week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Extended-Release Naltrexone | Buprenorphine-Naloxone
Number analyzed (Participants) | 283 | 287
Participants | 20 | 20

55. Secondary Outcome: Other Drug Use Over Time, Cocaine, W0
Description: Other drug use over time measuring cocaine at week 0
Time Frame: week 0
Measure: Count of Participants; unit: Participants
Arm/Group | Extended-Release Naltrexone | Buprenorphine-Naloxone
Number analyzed (Participants) | 283 | 287
Participants | 61 | 80

56. Secondary Outcome: Other Drug Use Over Time, Cocaine, W24
Description: Other drug use over time measuring cocaine at week 0
Time Frame: week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Extended-Release Naltrexone | Buprenorphine-Naloxone
Number analyzed (Participants) | 283 | 287
Participants | 5 | 2

57. Secondary Outcome: Other Drug Use Over Time, Stimulant, W0
Description: Other drug use over time measuring stimulant (cocaine, crack and amphetamine) at week 0
Time Frame: week 0
Measure: Count of Participants; unit: Participants
Arm/Group | Extended-Release Naltrexone | Buprenorphine-Naloxone
Number analyzed (Participants) | 283 | 287
Participants | 132 | 166

58. Secondary Outcome: Other Drug Use Over Time, Stimulant, W24
Description: Other drug use over time measuring stimulant (cocaine, crack and amphetamine) at week 24
Time Frame: week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Extended-Release Naltrexone | Buprenorphine-Naloxone
Number analyzed (Participants) | 283 | 287
Participants | 5 | 3

ADVERSE EVENTS:
Time Frame: Weeks 0-36
Description: Treatment emergent adverse events are those that occurred after study day of induction for those participants were inducted onto study medication.
Arm/Group | Extended-Release Naltrexone | Buprenorphine-Naloxone
All-Cause Mortality (participants affected / at risk) | 3/283 | 4/287
Serious Adverse Events (participants affected / at risk) | 41/283 | 31/287
Other Adverse Events (participants affected / at risk) | 118/283 | 135/287
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Extended-Release Naltrexone (N=283) | Buprenorphine-Naloxone (N=287)
Psychiatric (Psychiatric disorders) | 10 | 12
Infections and infestations (Infections and infestations) | 7 | 6
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1/270
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 17 | 8/270
General disorders and administration site conditions (General disorders) | 2 | 2/270
Gastrointestinal disorders (Gastrointestinal disorders) | 1 | 2/270
Respiratory, thoracic, and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 5 | 0/270
Nervous system disorders (Nervous system disorders) | 2 | 2/270
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 0 | 1/270
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 1 | 0/270
Hepatobiliary disorders (Hepatobiliary disorders) | 0 | 1/270
Eye disorders (Eye disorders) | 1 | 0/270
Reproductive system and breast disorders (Reproductive system and breast disorders) | 1 | 0/270
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Extended-Release Naltrexone (N=283) | Buprenorphine-Naloxone (N=287)
Gastrointestinal (Gastrointestinal disorders) | 36 | 58
Psychiatric (Psychiatric disorders) | 29 | 22
Injury poisoning and procedural complications (Injury, poisoning and procedural complications) | 18 | 22
Infections and infestations (Infections and infestations) | 22 | 22
Nervous system disorders (Nervous system disorders) | 29 | 27
General Disorders and Administration Site Conditions (General disorders) | 10 | 21
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 16 | 15
Investigations (Investigations) | 10 | 11
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 7 | 7
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 9 | 7
Metabolism and nutrition (Metabolism and nutrition disorders) | 6 | 4
Eye disorders (Eye disorders) | 6 | 3
Renal and urinary disorders (Renal and urinary disorders) | 4 | 5
Vascular disorders (Vascular disorders) | 1 | 6
Reproductive system and breast disorders (Reproductive system and breast disorders) | 2 | 3
Surgical and medical procedures (Surgical and medical procedures) | 0 | 3
Hepatbiliary disorders (Hepatobiliary disorders) | 1 | 1
Ear and labyrinth disorders (Ear and labyrinth disorders) | 1 | 1
Immune system disorders (Immune system disorders) | 0 | 1
Cardiac disorders (Cardiac disorders) | 1 | 0
Social circumstances (Social circumstances) | 1 | 0
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 1 | 0
Product issues (Product Issues) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-08-31): https://cdn.clinicaltrials.gov/large-docs/33/NCT02032433/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-27): https://cdn.clinicaltrials.gov/large-docs/33/NCT02032433/SAP_001.pdf